CLINICAL TRIAL: NCT01417858
Title: Short-term Intraocular Pressure Control After YAG Iridotomy - Comparison Between Brimonidine 0.1% vs. 0.2%
Brief Title: Intraocular Pressure Control After Anterior Segment Laser - Comparison Between 2 Drugs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Paraná (Other)
Responsible Party: Lucas Shiokawa, Universidade Federal do Parana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0299.0.208.000-10; 2376.270/2010-11 (Other: Hospital de Clinicas - UFPR - Research Ethics Committee)
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-06

CONDITIONS: Glaucoma, Narrow Angle
Keywords: intra-ocular pressure; iridectomy; gonioscopy; ocular tonometry
MeSH Terms: conditions — Glaucoma, Angle-Closure | interventions — Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- brimonidine 0.2% (Active Comparator)
  Interventions: Procedure: YAG laser peripheral iridotomy
- brimonidine 0.1% (Active Comparator)
  Interventions: Procedure: YAG laser peripheral iridotomy

INTERVENTIONS:
Procedure: YAG laser peripheral iridotomy — 1 drop 30 minutes before yag laser iridotomy
  Other Names: Alphagan
  Arms: brimonidine 0.2%
Procedure: YAG laser peripheral iridotomy — 1 drop 30 minutes before yag laser iridotomy
  Other Names: Alphagan z
  Arms: brimonidine 0.1%

SUMMARY:
The purpose of this study is to compare the intra-ocular (IOP) control efficacy between brimonidine 0.1% vs. 0.2% after laser peripheral iridotomy (LPI).

DETAILED DESCRIPTION:
Postoperative IOP elevation is one of the most common complications after LPI.Previous studies showed that brimonidine 0.2% is effective in blunting IOP spikes after LPI.This prospective randomized double-masked interventional study will include patients with bilateral narrow angles, defined by irido-trabecular contact in >180o on gonioscopy.Pilocarpine 1% will be used in both eyes, and 30 minutes later, brimonidine 0.1% randomly used in one eye and brimonidine 0.2% in the contra-lateral eye. LPI with Nd:YAG laser is performed 30 minutes later in both eyes by a single glaucoma specialist. IOP measurements are assessed before the use of any eyedrop (basal IOP), 30 minutes after pilocarpine (pre-brimonidine), and 30, 60, 120, 180 minutes after LPI. Pachymetry, ultrasonic biometry, gonioscopy, and total YAG laser energy are recorded. Non-parametric test will be used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* bilateral narrow angles, defined by irido-trabecular contact in >180o on gonioscopy

Exclusion Criteria:

* previous cataract surgery

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-12 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
intra-ocular pressure increase | one year
  mean intra-ocular pressure increase after laser peripheral iridotomy

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Shiokawa, MD, Principal Investigator — Universidade Federal do Parana
Locations (1):
- Universidade Federal do Parana, Curitiba, Paraná, Brazil

REFERENCES:
- [Background] Brazier DJ. Neodymium-YAG laser iridotomy. J R Soc Med. 1986 Nov;79(11):658-60. doi: 10.1177/014107688607901115. PMID 3795210
- [Background] Chen TC, Ang RT, Grosskreutz CL, Pasquale LR, Fan JT. Brimonidine 0.2% versus apraclonidine 0.5% for prevention of intraocular pressure elevations after anterior segment laser surgery. Ophthalmology. 2001 Jun;108(6):1033-8. doi: 10.1016/s0161-6420(01)00545-0. PMID 11382625
- [Background] Chen TC. Brimonidine 0.15% versus apraclonidine 0.5% for prevention of intraocular pressure elevation after anterior segment laser surgery. J Cataract Refract Surg. 2005 Sep;31(9):1707-12. doi: 10.1016/j.jcrs.2005.02.035. PMID 16246772
- [Background] Drake MV. Neodymium:YAG laser iridotomy. Surv Ophthalmol. 1987 Nov-Dec;32(3):171-7. doi: 10.1016/0039-6257(87)90092-0. PMID 3328316
- [Background] Hartenbaum D, Wilson H, Maloney S, Vacarelli L, Orillac R, Sharpe E. A randomized study of dorzolamide in the prevention of elevated intraocular pressure after anterior segment laser surgery. Dorzolamide Laser Study Group. J Glaucoma. 1999 Aug;8(4):273-5. PMID 10464738
- [Background] Kashiwagi K, Abe K, Tsukahara S. Quantitative evaluation of changes in anterior segment biometry by peripheral laser iridotomy using newly developed scanning peripheral anterior chamber depth analyser. Br J Ophthalmol. 2004 Aug;88(8):1036-41. doi: 10.1136/bjo.2003.036715. PMID 15258021
- [Background] Khodadoust AA, Arkfeld DF, Caprioli J, Sears ML. Ocular effect of neodymium-YAG laser. Am J Ophthalmol. 1984 Aug 15;98(2):144-52. doi: 10.1016/0002-9394(87)90348-5. PMID 6548087
- [Background] Robin AL, Arkell S, Gilbert SM, Goossens AA, Werner RP, Korshin OM. Q-switched neodymium-YAG laser iridotomy. A field trial with a portable laser system. Arch Ophthalmol. 1986 Apr;104(4):526-30. doi: 10.1001/archopht.1986.01050160082017. PMID 3513746
- [Background] Schrems W, Eichelbronner O, Krieglstein GK. The immediate IOP response of Nd-YAG-laser iridotomy and its prophylactic treatability. Acta Ophthalmol (Copenh). 1984 Oct;62(5):673-80. doi: 10.1111/j.1755-3768.1984.tb05794.x. PMID 6548856
- [Background] Wetzel W. Ocular aqueous humor dynamics after photodisruptive laser surgery procedures. Ophthalmic Surg. 1994 May;25(5):298-302. PMID 8058261